CLINICAL TRIAL: NCT05394987
Title: Spectacle Correction for the Treatment of Amblyopia
Brief Title: Optical Correction and Visual Functions of Adults With Amblyopia
Acronym: SPECTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Eye and Vision Research (Other)
Collaborators: The Hong Kong Polytechnic University (Other); University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPECTRA
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Amblyopia
Keywords: Amblyopia; Binocular vision; Suppression; Plasticity; Optical correction
MeSH Terms: conditions — Amblyopia | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: Within-subject, pre-post interventional study, measuring the effect of optical correction on visual function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optical correction (Experimental): Prescription of spectacles for full-time wear to correct refractive error
  Interventions: Device: Spectacles

INTERVENTIONS:
Device: Spectacles — Prescription of refractive error correction in spectacles. Refractive error to be determined as part of standard optometric eye exam (performed by registered optometrist).
  Guidelines for optical correction for the prescription of the study spectacles (based on Pediatric Eye Disease Investigator Group [PEDIG] amblyopia clinical trial protocols): Hypermetropia: not undercorrected by >+1.50D spherical equivalent and the reduction in plus sphere must be identical between the two eyes. Anisometropia: full correction of the anisometropic difference. Astigmatism: cylinder power in each eye should be within ≤±0.50D of fully correcting the astigmatism for each eye. If cylinder power is ≥1.00D, the prescribed axis in both eyes should be within ≤±6 deg of the cycloplegic refraction axis.
  Appropriate refractive error correction will be prescribed. Participants will be instructed to wear the optical correction full-time (i.e., >50% of waking hours) for the duration of the study.

SUMMARY:
Amblyopia is a developmental anomaly resulting from abnormal visual experiences in early life. Amblyopia causes reduced visual acuity in the absence of a pathology. Adult sensory systems are believed to be structurally invariant beyond early, critical periods of development. However, recent evidence suggest that visual functions in adults with amblyopia can be improved with optical correction alone. This study aims to investigate whether improvements in best corrected visual acuity and other visual functions can result following appropriate optical correction in adults with amblyopia. Functional measures relating to vision, binocular vision, and eye movements will be used to assess the efficacy of refractive correction for improving vision. This study will help us better understand the improvements in visual functions following optical correction, as well as the mechanisms underlying neuroplasticity in adults with amblyopia.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 (inclusive) years of age
* Anisometropic amblyopia (difference of ≥0.50D spherical equivalent or ≥1.50D astigmatism between eyes) or mixed mechanism amblyopia (strabismus and anisometropia)
* Best corrected visual acuity (BCVA) in the amblyopic eye of 0.3 logMAR to 1.0 logMAR (inclusive)
* BCVA in the non-amblyopic eye of 0.1 logMAR or better, and an interocular VA difference of 2 logMAR lines or more
* Difference of 1.00D or more between current refractive correction and study prescription
* Good general health

Exclusion Criteria:

* Other pathological ocular anomalies known to cause reduced visual acuity
* Presbyopia (based on amplitude of accommodation)
* Inability to tolerate prescribed refractive correction in spectacles (e.g., due to aniseikonia)
* Contraindication to cycloplegic eye drops
* Currently under amblyopia treatment/therapy
* Inability to comprehend test instructions and/or provide consent
* Eccentric fixation
* >-6.00DS of myopia in either eye with spectacles
* Bilateral amblyopia
* Presence of amblyopia that is not due to strabismus and/or anisometropia
* Presence of (current or previous) psychiatric, visual, or neurological disorders

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity of the amblyopic eye pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  The size of the smallest line of letters read accurately on an ETDRS chart.
Best corrected visual acuity of the amblyopic eye post-intervention | Approx. 5 mins, on completion of study (week 24)
  The size of the smallest line of letters read accurately on an ETDRS chart.

SECONDARY OUTCOMES:
Best corrected visual acuity of the amblyopic eye during intervention | Approx. 5 mins, every 4 weeks from start of intervention
  The size of the smallest line of letters read accurately on an ETDRS chart.
Fellow eye distance visual acuity pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  The size of the smallest line of letters read accurately on an ETDRS chart.
Fellow eye distance visual acuity post-intervention | Approx. 5 mins, on completion of study (week 24)
  The size of the smallest line of letters read accurately on an ETDRS chart.
Fellow eye distance visual acuity during-intervention | Approx. 5 mins, every 4 weeks from start of intervention
  The size of the smallest line of letters read accurately on an ETDRS chart.
Binocular distance visual acuity pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  The size of the smallest line of letters read accurately on an ETDRS chart.
Binocular distance visual acuity post-intervention | Approx. 5 mins, on completion of study (week 24)
  The size of the smallest line of letters read accurately on an ETDRS chart.
Binocular distance visual acuity during intervention | Approx. 5 mins, every 4 weeks from start of intervention
  The size of the smallest line of letters read accurately on an ETDRS chart.
Near visual acuity of amblyopic eye pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Near visual acuity of amblyopic eye post-intervention | Approx. 5 mins, on completion of study (week 24)
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Near visual acuity of amblyopic eye during intervention | Approx. 5 mins,every 4 weeks from start of intervention
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Near visual acuity of fellow eye pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Near visual acuity of fellow eye post-intervention | Approx. 5 mins, on completion of study (week 24)
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Near visual acuity of fellow eye during intervention | Approx. 5 mins, every 4 weeks from start of intervention
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Near binocular visual acuity pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Near binocular visual acuity post-intervention | Approx. 5 mins, on completion of study (week 24)
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Near binocular visual acuity during intervention | Approx. 5 mins, every 4 weeks from start of intervention
  The size of the smallest line of letters read accurately on a near ETDRS chart.
Amblyopic eye contrast sensitivity pre-intervention | Approx. 10 mins, baseline (day 1 of spectacle wear)
  Computer-based measurement of contrast sensitivity
Amblyopic eye contrast sensitivity post-intervention | Approx. 10 mins, on completion of study (week 24)
  Computer-based measurement of contrast sensitivity
Amblyopic eye contrast sensitivity during intervention | Approx. 10 mins, every 4 weeks from start of intervention
  Computer-based measurement of contrast sensitivity
Stereopsis pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  Smallest disparity on the Randot preschool test reported accurately.
Stereopsis post-intervention | Approx. 5 mins, on completion of study (week 24)
  Smallest disparity on the Randot preschool test reported accurately.
Stereopsis during intervention | Approx. 5 mins, every 4 weeks from start of intervention
  Smallest disparity on the Randot preschool test reported accurately.
Angle of strabismus pre-intervention | Approx. 5 mins,baseline (day 1 of spectacle wear)
  Prismatic power required to neutralise the angle of deviation on alternating prism cover test.
Angle of strabismus post-intervention | Approx. 5 mins, on completion of study (week 24)
  Prismatic power required to neutralise the angle of deviation on alternating prism cover test.
Angle of strabismus during intervention | Approx. 5 mins, every 4 weeks from start of intervention
  Prismatic power required to neutralise the angle of deviation on alternating prism cover test.
Amblyopic eye fixation stability pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  Eye position recorded with high-speed eye tracker during fixation as quantified by bivariate contour ellipse area (BCEA).
Amblyopic eye fixation stability post-intervention | Approx. 5 mins, on completion of study (week 24)
  Eye position recorded with high-speed eye tracker during fixation as quantified by bivariate contour ellipse area (BCEA).
Amblyopic eye fixation stability during intervention | Approx. 5 mins, every 4 weeks from start of intervention
  Eye position recorded with high-speed eye tracker during fixation as quantified by bivariate contour ellipse area (BCEA).
Fellow (non-amblyopic) eye fixation stability pre-intervention | Approx. 5 mins, baseline (day 1 of spectacle wear)
  Eye position recorded with high-speed eye tracker during fixation as quantified by bivariate contour ellipse area (BCEA).
Fellow (non-amblyopic) eye fixation stability post-intervention | Approx. 5 mins, on completion of study (week 24)
  Eye position recorded with high-speed eye tracker during fixation as quantified by bivariate contour ellipse area (BCEA).
Fellow (non-amblyopic) eye fixation stability during intervention | Approx. 5 mins, every 4 weeks from start of intervention
  Eye position recorded with high-speed eye tracker during fixation as quantified by bivariate contour ellipse area (BCEA).
Interocular suppression pre-intervention | Approx. 10 mins, baseline (day 1 of spectacle wear)
  Computer-based measurement of interocular suppression.
Interocular suppression post-intervention | Approx. 10 mins, on completion of study (week 24)
  Computer-based measurement of interocular suppression.
Interocular suppression during intervention | Approx. 10 mins, every 4 weeks from start of intervention
  Computer-based measurement of interocular suppression.
Quality of life pre-intervention | Approx.15-20 mins, baseline (day 1 of spectacle wear)
  Questionnaire scores for:
  1. Amblyopia and Strabismus Questionnaire
  2. World Health Organization Quality of Life-BREF
Quality of life post-intervention | Approx. 15-20 mins, on completion of study (week 24)
  Questionnaire scores for:
  1. Amblyopia and Strabismus Questionnaire
  2. World Health Organization Quality of Life-BREF

OTHER OUTCOMES:
Electrical potentials pre-intervention | Approx. 60 mins, baseline (day 1 of spectacle wear)
  Electroencephalography (EEG) measures:
  Visual evoked potentials for high and low contrast stimuli (monocular: fellow eye and amblyopic eye)
Electrical potentials post-intervention | Approx. 60 mins, on completion of study (week 24)
  Electroencephalography (EEG) measures:
  Visual evoked potentials for high and low contrast stimuli (monocular: fellow eye and amblyopic eye)
Electrical potentials during intervention | Approx. 60 mins, 12 weeks from baseline (day 1 of spectacle wear)
  Electroencephalography (EEG) measures:
  Visual evoked potentials for high and low contrast stimuli (monocular: fellow eye and amblyopic eye)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Thompson, PhD, Principal Investigator — Centre for Eye and Vision Research Limited; Ken WS Tan, PhD, Study Director — Centre for Eye and Vision Research Limited
Locations (2):
- University of Waterloo, Waterloo, Ontario, Canada
- Centre for Eye and Vision Research Limited, Hong Kong, Guangdong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared on request
Supporting Information: Study Protocol, SAP
Time Frame: After publication of study results for an indefinite period.
Access Criteria: Upon reasonable request and approved by the study principal investigator.

REFERENCES:
- [Derived] Tan KWS, Park ASY, Cheung BWS, Wong GHT, Thompson B; SPECTRA study team. SPEctacle Correction for the TReatment of Amblyopia (SPECTRA): study protocol for a prospective non-randomised interventional trial in adults with anisometropic/mixed mechanism amblyopia. BMJ Open. 2024 Jul 1;14(6):e080151. doi: 10.1136/bmjopen-2023-080151. PMID 38950991